CLINICAL TRIAL: NCT04182672
Title: Study to Assess the Safety and Efficacy of FX006 Administered to Patients With Greater Trochanteric Bursitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Pacira Pharmaceuticals, Inc (Industry)
Responsible Party: Principal Investigator, Pritish Bawa, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSC-MS-18-0672
Record Dates: First submitted 2019-11-27; First posted 2019-12-02 (Actual); Results first posted 2024-01-02 (Actual); Last update posted 2024-01-02 (Actual); Status verified 2023-12

CONDITIONS: Trochanteric Bursitis
Keywords: Hip bursitis; hip pain
MeSH Terms: interventions — FX006

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- FX006 (Experimental)
  Interventions: Drug: FX006

INTERVENTIONS:
Drug: FX006 — Subjects will be injected with the 5mL of FX006. This injection may be followed with up to 3mL of ropivacaine (depending on the capacity of the bursa), under ultrasound guidance.

SUMMARY:
The purpose of this study is to determine the safety and efficacy of FX006 in bursal injections and to assess the patient's impression to change in their chronic pain, following treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written consent to participate in the study
* Symptoms consistent with greater trochanteric bursitis for greater than or equal to 3 months prior to screening (patient reported is acceptable)
* Pain in hip for greater than 15 days over the last month (as reported by the patient).
* Hip bursitis as determined by clinical examination and clinical features. Where Magnetic Resonance Imaging (MRI) data is available, it will be used to confirm the bursitis diagnosis. Also, pain relief in subjects that have been treated with bursal injections containing an anesthetic (such as ropivacaine) is in itself indicative of bursitis.
* Body mass index (BMI) less than or equal to 40 kg/m2
* Ambulatory and in good general health
* Willing and able to comply with the study procedures and visit schedules and able to follow verbal and written instructions.
* Willing to abstain from use of protocol-restricted medications during the study

Exclusion Criteria:

* Hip Arthroplasty
* Hip osteoarthritis, iliopsoas bursitis, reactive arthritis,rheumatoid arthritis, psoriatic arthritis, ankylosing spondylitis, or arthritis associated with inflammatory bowel disease
* History of local infection around the bursa.
* Lack of pain relief with the intrabursal treatments containing an anesthetic
* Intra-bursal treatment of any bursa with any of the following agents within three (3) months of screening: any corticosteroid preparation (investigational or marketed, including FX006); and/or six (6) months for any biologic agent (e.g., platelet rich plasma (PRP) injection, stem cells, prolotherapy, amniotic fluid injection; investigational or marketed).
* Parenteral or oral corticosteroids (investigational or marketed) within 3 months of Screening
* Inhaled, intranasal or topical corticosteroids (investigational or marketed) within 2 weeks of screening.
* Females who are pregnant or nursing or plan to become pregnant during the study; women who plan to conceive

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2020-08-12 (Actual); Primary Completion 2022-12-14 (Actual); Study Completion 2022-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pritish Bawa, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Units Other Than Participants: hips
Period: Overall Study
Arm/Group | FX006
Started | 22; 24 hips
Completed | 22; 24 hips
Not Completed | 0; 0 hips

BASELINE CHARACTERISTICS:
Arm/Group | FX006
Number analyzed (Participants) | 22
Age, Continuous [Median (Full Range); unit: years] | 62.5 [40 to 76]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 6
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 7
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 12
  More than one race | 0
  Unknown or Not Reported | 7
Region of Enrollment [Number; unit: participants]
  United States | 22
Baseline Numeric Pain Rating Scale (NPRS) Score [Median (Full Range); unit: score on a scale] — Numeric Pain Rating Scale total score ranges from 0 (no pain) to 10 (most intense pain imaginable).
  score on a scale | 5 [2 to 10]
Baseline Patient Global Impression of Change (PGIC) score [Median (Full Range); unit: score on a scale] — The PGIC is a 7 point scale ranging from very much improved (1) to very much worsened (7)
  score on a scale | 2 [1 to 4]

OUTCOME MEASURES:

1. Primary Outcome: Change in Pain From Baseline as Assessed by the Numeric Pain Rating Scale (NPRS) Score
Description: Numeric Pain Rating Scale total score ranges from 0 (no pain) to 10 (most intense pain imaginable).
Time Frame: Baseline,week 12
Population: Data were not collected for two participants in the FX006 arm.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | FX006
Number analyzed (Participants) | 20
score on a scale | -2.25 (3.64)

2. Secondary Outcome: Patient Global Impression of Change (PGIC) Score
Description: The PGIC is a 7 point scale ranging from very much improved (1) to very much worsened (7)
  1. No change (or condition has got worse)
  2. Almost the same, hardly any change at all
  3. A little better, but no noticeable change
  4. Somewhat better, but the change has not made any real difference
  5. Moderately better, and a slight but noticeable change
  6. Better, and a definite improvement that has made a real and worthwhile difference
  7. A great deal better, and a considerable improvement that has made all the difference
Time Frame: from start of treatment to week 12 of treatment
Population: Data were not collected for two participants in the FX006 arm.
Measure: Median (Full Range); unit: score on a scale
Arm/Group | FX006
Number analyzed (Participants) | 20
score on a scale | 5 [1 to 7]

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | FX006
All-Cause Mortality (participants affected / at risk) | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22
Other Adverse Events (participants affected / at risk) | 6/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FX006 (N=22)
Hip Pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Fall (Nervous system disorders) | 1 (1)
Pain at Injection Site (Musculoskeletal and connective tissue disorders) | 4 (4)
Subcutaneous and Skin Disorders-other-lump at injection site (Musculoskeletal and connective tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
Adverse event relating to fall was not related to the treatment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-02-12): https://cdn.clinicaltrials.gov/large-docs/72/NCT04182672/Prot_SAP_000.pdf